CLINICAL TRIAL: NCT03673111
Title: A Randomised, Placebo Controlled First in Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Y14 in Adult Subjects
Brief Title: Study of the Gut Hormone Analogue Y14 in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ICIM/2016/Y14/01; 2017-000380-33 (EudraCT Number)
Record Dates: First submitted 2018-05-23; First posted 2018-09-17 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- 1.0 mg Y14 (A1) (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 2.0 mg Y14 (A1) (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 6.0 mg Y14 (A1) (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 9.0 mg Y14 (A2) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 18.0 mg Y14 (A5) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 36.0 mg Y14 (A6) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- Placebo (B) (Placebo Comparator): 5 subcutaneous injections of 0.9% saline, over a 4 week treatment period
  Interventions: Drug: Placebo
- 9-26.0 mg (B1) (Experimental): Y14 multiple dose, subcutaneous 5 doses over a 4 week treatment period: escalating doses to a max of 26 mg
  Interventions: Drug: Y14
- 9-36 mg (B2) (Experimental): Y14 multiple dose, subcutaneous 4 doses over a 4 week treatment period: escalating doses to a max of 36 mg
  Interventions: Drug: Y14
- 12-36 mg (B3) (Experimental): Y14 multiple dose, subcutaneous 4 doses over a 4 week treatment period: escalating doses to a max of 36 mg
  Interventions: Drug: Y14
- Placebo (A) (Placebo Comparator): Single subcutaneous injection of 0.9% saline
  Interventions: Drug: Placebo
- 9 mg Y14 (A3) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 9 mg Y14 (A4) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 18 mg Y14 (A7) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 36 mg Y14 (A8) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14
- 36 mg Y14 (A9) with varied formulation (Experimental): Y14 single dose, subcutaneous
  Interventions: Drug: Y14

INTERVENTIONS:
Drug: Y14 — Gut hormone analogue
  Other Names: Gut hormone analogue
  Arms: 1.0 mg Y14 (A1); 12-36 mg (B3); 18 mg Y14 (A7) with varied formulation; 18.0 mg Y14 (A5) with varied formulation; 2.0 mg Y14 (A1); 36 mg Y14 (A8) with varied formulation; 36 mg Y14 (A9) with varied formulation; 36.0 mg Y14 (A6) with varied formulation; 6.0 mg Y14 (A1); 9 mg Y14 (A3) with varied formulation; 9 mg Y14 (A4) with varied formulation; 9-26.0 mg (B1); 9-36 mg (B2); 9.0 mg Y14 (A2) with varied formulation
Drug: Placebo — 0.9% saline
  Other Names: Saline
  Arms: Placebo (A); Placebo (B)

SUMMARY:
A randomised, placebo controlled Phase I study to investigate investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of Y14 in adult subjects.

DETAILED DESCRIPTION:
Objectives:

Primary Objective

* To investigate the safety and tolerability of single doses of Y14 in overweight/obese but otherwise healthy male subjects.
* To investigate the safety and tolerability of multiple doses of Y14 in overweight/obese male subjects with normal glucose tolerance, Type 2 diabetes or prediabetes.

Secondary Objectives

* To assess the pharmacokinetic (PK) profile of single doses of Y14 in overweight/obese but otherwise healthy male subjects.
* To assess the PK profile of multiple ascending doses of Y14 in overweight/obese male subjects with normal glucose tolerance, Type 2 diabetes or prediabetes.

Exploratory Objective

* To investigate the effects of multiple doses of Y14 on food consumption, body weight and glucose tolerance in overweight/obese male subjects with normal glucose tolerance, Type 2 diabetes or prediabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18 to 65 years inclusive with BMI between 25.0 and 38.0 kg/m2 inclusive;
2. (PART B only) Subjects who have normal glucose tolerance, Type 2 diabetes, impaired glucose tolerance or impaired fasting glucose according to WHO 2006 and 2011 criteria;
3. Subjects who are otherwise healthy enough to participate, as determined by pre-study medical history, physical examination and 12-lead ECG;
4. Subjects whose clinical laboratory test results are either within the normal range or if outside this range the abnormalities are judged to be not clinically relevant and are acceptable to the Investigator;
5. Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening;
6. Subjects who are negative for drugs of abuse and alcohol tests at screening and admissions;
7. Subjects who are non-smokers for at least 3 months preceding screening;
8. Subjects who agree to use medically acceptable methods of contraception for at least 3 months after study drug administration;
9. Subjects who agree not to donate sperm for at least 3 months after study drug administration;
10. Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

1. Subjects who do not conform to the above inclusion criteria;
2. Subjects who have a clinically relevant history or presence of gastrointestinal (especially associated with vomiting), respiratory, renal, hepatic, haematological, lymphatic, neurological (especially if associated with balance disorders or vomiting e.g. migraine or labyrinthitis), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders;
3. Subjects who have a clinically relevant surgical history;
4. Subjects who are currently taking any of the following classes of diabetes medications: thiazolidinediones, dipeptidyl peptidase IV inhibitors ('gliptins'), GLP-1 analogues, and insulin;
5. Subjects who have a history of relevant and severe atopy e.g. asthma, angioedema requiring emergency treatment, severe hayfever requiring regular treatment (i.e. taking antihistamines and/or glucocorticoids more regularly than 3 times a week), severe eczema requiring regular treatment (i.e. taking antihistamines and/or glucocorticoids more regularly than 3 times a week);
6. Subjects who have a history of relevant drug hypersensitivity;
7. Subjects who have a history of alcohol abuse or alcohol dependence according to DSMIV criteria within the last 2 years;
8. Subjects who have a history of drug or substance abuse according to DSM-IV criteria within the last 2 years;
9. Subjects who have a history of clinically significant migraine as judged by the Investigator. Subjects can be included if they have not had a migraine for the last 3 years;
10. Subjects with a history of pancreatitis or pancreatic cancer;
11. Subjects who consume more than 21 units of alcohol a week (unit = 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer);
12. Subjects who have a significant infection or known inflammatory process on screening;
13. Subjects who have acute gastrointestinal symptoms at the time of screening or admission (e.g. nausea, vomiting, diarrhoea, heartburn);
14. Subjects who have an acute infection such as influenza at the time of screening or admission;
15. Subjects who have used prescription drugs within 2 weeks of first dosing. For Part B, patients are allowed to be treated for their diabetes with monotherapy with a sulphonylurea, metformin, or a SGLT-2 inhibitor, dual therapy with any two of the following drug types: a sulphonylurea, metformin, and/or a SGLT-2 inhibitor; triple therapy with a sulphonylurea, metformin, and a SGLT-2 inhibitor. In addition patients in Part B are allowed to take hypolipidaemic and/or antihypertensive treatments, provided that the doses have not been altered within the 4 weeks prior to entering the study. Other medications may be allowed if the Investigator and Sponsor both agree that they will not affect the outcome of the study or the safety of the subject.
16. Subjects who have used over the counter medication excluding routine vitamins and paracetamol but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first dosing, unless agreed as not clinically relevant by the Principal Investigator and Sponsor;
17. Subjects who have donated blood within 3 months prior to screening; Subjects who have donated plasma within the 7 days prior to screening; Subjects who have donated platelets within the 6 weeks prior to screening
18. Subjects who have used any investigational drug in any clinical trial within 3 months of their first admission date;
19. Subjects who have received the last dose of investigational drug greater than 3 months ago but who are on extended follow-up;
20. Subjects who have previously received Y14;
21. Subjects who are vegans, vegetarian or have any dietary restriction (unless agreed as not clinically relevant by the PI and Sponsors);
22. Subjects who cannot communicate reliably with the Investigator;
23. Subjects who are unlikely to co-operate with the requirements of the study;
24. History or evidence of abnormal eating behaviour, as observed through the Dutch Eating Behaviour (DEBQ) and SCOFF questionnaires at screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bloom, FMedSci, FRS, Study Director — Sponsor Chief Investigator, Imperial College London
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan TM, Minnion J, Khoo B, Ball LJ, Malviya R, Day E, Fiorentino F, Brindley C, Bush J, Bloom SR. Safety and efficacy of an extended-release peptide YY analogue for obesity: A randomized, placebo-controlled, phase 1 trial. Diabetes Obes Metab. 2021 Jul;23(7):1471-1483. doi: 10.1111/dom.14358. Epub 2021 Mar 9. PMID 33606914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single ascending dose - Part A: Cohort A1 comprised 4 subjects (3 active and 1 placebo): each volunteer was dosed in three treatment periods (TP) with three ascending dose levels (doses 1 mg, 2 mg, 6 mg Y14), with minimum washouts of 1 week between Day 1 of each TP. Within each TP three subjects were given the study drug and one placebo (sterile 0.9% [w/v] saline. Each volunteer in Cohort A2 onwards was dosed only once.
  Multiple ascending dose - Part B: Each participant received up to 5 doses
Groups:
- Y14 Single Ascending Dose (A1: TP1, TP2 & TP3): Sequential cross-over group received either Saline or 1 mg dose Y14 (A1) single dose, subcutaneous injection in the first treatment period; Saline or 2 mg dose Y14 single dose, subcutaneous injection in the second period, Saline or 6 mg dose Y14 single dose, subcutaneous injection in the third treatment period.
  Treatment periods were 12-15 days apart.
- 9.0 mg (A2); 9 mg (A3); 9 mg (A4); 18.0 mg (A5); 36.0 mg (A6); 18 mg (A7); 36 mg (A8); 36 mg (A9): Y14 single dose, subcutaneous
  Y14: Gut hormone analogue
- Placebo SAD (A2-A9): 0.9% saline
  Placebo: 0.9% saline
- Placebo (Part B): 0.9% saline multiple subcutaneous injection:
  5 injections over a 4 week treatment period
- 9-26.0 mg (B1): Y14 multiple dose, subcutaneous 5 doses over a 4 week treatment period: escalating doses up to maximum 26 mg
  Y14: Gut hormone analogue
- 9-36 mg (B2): Y14 multiple dose, subcutaneous 4 doses over a 4 week treatment period: escalating doses up to maximum 36 mg
  Y14: Gut hormone analogue
- 12-36 mg (B3): Y14 multiple dose, subcutaneous 4 doses over a 4 week treatment period: escalating doses up to a maximum of 36 mg
  Y14: Gut hormone analogue
Period: Overall Study
Arm/Group | Y14 Single Ascending Dose (A1: TP1, TP2 & TP3) | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD (A2-A9) | Placebo (Part B) | 9-26.0 mg (B1) | 9-36 mg (B2) | 12-36 mg (B3)
Started (One participant was withdrawn after treatment period 2 and a replacement subject was recruited for treatment period 3) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6
Completed (One participant was withdrawn after treatment period 2 and a replacement subject was recruited for treatment period 3) | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAD A1: Sequential cross-over group received either Saline or 1 mg dose Y14 (A1) single dose, subcutaneous injection in the first treatment period; Saline or 2 mg dose Y14 single dose, subcutaneous injection in the second period, Saline or 6 mg dose Y14 single dose, subcutaneous injection in the third treatment period. Treatment periods were 12-15 days apart.
- Placebo SAD A2-A9: 0.9% saline
  Placebo: 0.9% saline
- 9-26.0 mg (B1): Y14 multiple dose, subcutaneous 5 doses over a 4 week treatment period: escalating dose up to 26 mg
  Y14: Gut hormone analogue
- 9-36 mg (B2): Y14 multiple dose, subcutaneous 5 doses over a 4 week treatment period: escalating dose up to 36 mg
  Y14: Gut hormone analogue
- 12-36 mg (B3): Y14 multiple dose, subcutaneous 5 doses over a 4 week treatment period: escalating dose up to 36 mg.
  Y14: Gut hormone analogue
- Total: Total of all reporting groups
Arm/Group | SAD A1 | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD A2-A9 | Placebo (Part B) | 9-26.0 mg (B1) | 9-36 mg (B2) | 12-36 mg (B3) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.44) | 28.2 (5.02) | 47.8 (10.8) | 41.2 (13.3) | 45.6 (14.9) | 47.8 (1.5) | 40.4 (13.3) | 44.2 (12.5) | 37.0 (12.2) | 44.8 (11.5) | 49.5 (11.9) | 36.7 (10.0) | 42.3 (9.6) | 40.8 (9.7) | 42.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 8
  White | 5 | 4 | 4 | 4 | 5 | 5 | 4 | 4 | 5 | 5 | 5 | 5 | 5 | 6 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 77
Body Weight (kg) [Mean (Standard Deviation); unit: kg] | 89.0 (12.41) | 101.6 (12.7) | 100.4 (11.3) | 86.2 (11.78) | 101.6 (9.6) | 93.3 (5.60) | 87.4 (13.3) | 92.4 (16.47) | 88.6 (7.4) | 97.5 (14.9) | 93.2 (14.8) | 97.5 (14.0) | 95.2 (9.8) | 92.0 (8.1) | 92.0 (12.09)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (2.05) | 30.0 (2.70) | 30.8 (1.9) | 27.6 (2.4) | 30.6 (1.8) | 28.8 (1.87) | 27.0 (2.9) | 30.6 (4.2) | 26.6 (0.9) | 30.1 (2.9) | 29.7 (3.1) | 30.2 (3.9) | 30.2 (2.9) | 29.5 (2.1) | 29.3 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (Safety and Tolerability)
Description: As assessed by reporting of adverse events, vital signs, physical examination, clinical laboratory safety assessments, and ECG parameters.
  Possibly or definitely related to study drug
Time Frame: Up to 73 days after dosing
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (A1): 0.9% saline single subcutaneous injection
- 1.0 mg (A1) TP1; 2.0 mg (A1) TP2; 6.0 mg (A1) TP3; 9 mg (A4); 9 mg (A3); 9.0 mg (A2); 18 mg (A7); 18.0 mg (A5); 36 mg (A8); 36.0 mg (A6); 36 mg (A9): Y14 single dose, subcutaneous
  Y14: Gut hormone analogue
- 9 mg Y14 (B1); 12 mg Y14 (B1); 16 mg Y14 (B1); 20 mg Y14 (B1); 26 mg Y14 (B1): Y14 multiple dose, subcutaneous injection:
  1 of 5 doses over a 4 week treatment period at escalating doses.
  Y14: Gut hormone analogue
- 9 mg Y14 (B2); 12 mg Y14 (B3); 24 mg Y14 (B2); 24 mg Y14 (B3); 36 mg Y14 (B2); 36 mg Y14 (B3): Y14 multiple dose, subcutaneous injection:
  1 of 4 doses over a 4 week treatment period at escalating doses.
  Y14: Gut hormone analogue
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | 9 mg (A4) | 9 mg (A3) | 9.0 mg (A2) | 18 mg (A7) | 18.0 mg (A5) | 36 mg (A8) | 36.0 mg (A6) | 36 mg (A9) | Placebo SAD A2-A9 | Placebo (Part B) | 9 mg Y14 (B1) | 9 mg Y14 (B2) | 12 mg Y14 (B1) | 12 mg Y14 (B3) | 16 mg Y14 (B1) | 20 mg Y14 (B1) | 24 mg Y14 (B2) | 24 mg Y14 (B3) | 26 mg Y14 (B1) | 36 mg Y14 (B2) | 36 mg Y14 (B3)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 1 | 1 | 3 | 5 | 4 | 1 | 5 | 5 | 4 | 5 | 5 | 3 | 3 | 5 | 4 | 6 | 5 | 6 | 6 | 6 | 5 | 6 | 5 | 6

2. Secondary Outcome: Cmax
Description: The maximum observed concentration
Time Frame: For Part A, Cohorts A3 to A9 - up to 840 hour post dose. For Part B - up to day 70 post 1st dose
Population: PK Parameters: N/A= For the doses given to cohorts A1, A2 and A3, Y14 was below the LLOQ(<0.2 ng/mL) in most samples (BLQ=below the limit of quantification), so the data for cohort A4 onwards are presented. Only subjects receiving Y14 were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 36 mg Y14 (B2) 1st Dose; 36mg Y14 (B2) 2nd Dose; 12 mg Y14 (B3); 24 mg Y14 (B3); 36 mg Y14 (B3) 1st Dose; 36 mg Y14 (B3) 2nd Dose: Y14 multiple dose, subcutaneous injection:
  1 of 4 doses over a 4 week treatment period at escalating doses.
  Y14: Gut hormone analogue
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD A2-A9 | Placebo (Part B) | 9 mg Y14 (B1) | 12 mg Y14 (B1) | 16 mg Y14 (B1) | 20 mg Y14 (B1) | 26 mg Y14 (B1) | 9 mg Y14 (B2) | 24 mg Y14 (B2) | 36 mg Y14 (B2) 1st Dose | 36mg Y14 (B2) 2nd Dose | 12 mg Y14 (B3) | 24 mg Y14 (B3) | 36 mg Y14 (B3) 1st Dose | 36 mg Y14 (B3) 2nd Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | 0.459 (44) | 0.383 (46) | 0.607 (111) | 0.677 (66) | 0.908 (81) | 0.704 (59) | NA (NA) — BLQ | NA (NA) — BLQ | 0.640 (39) | 0.870 (26) | 1.32 (35) | 1.64 (19) | 1.48 (49) | 0.389 (41) | 0.702 (52) | 1.4 (21) | 1.1 (66) | 0.355 (37) | 0.787 (35) | 1.35 (20) | 1.54 (41)

3. Secondary Outcome: AUC 0-72h
Description: The area under the concentration versus time curve from time zero to 72 h postdose, calculated by the mixed linear/log trapezoidal rule
Time Frame: Up to 72hr after dosing
Population: PK Parameters: N/A = For the doses given to cohorts A1, A2, A3 and A5, Y14 was below the LLOQ(<0.2 ng/mL) in most samples (BLQ=below the limit of quantification), so the data for cohort A4 and cohort A6 onwards are presented. Only subjects receiving Y14 were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD A2-A9 | Placebo (Part B) | 9 mg Y14 (B1) | 12 mg Y14 (B1) | 16 mg Y14 (B1) | 20 mg Y14 (B1) | 26 mg Y14 (B1) | 9 mg Y14 (B2) | 24 mg Y14 (B2) | 36 mg Y14 (B2) 1st Dose | 36mg Y14 (B2) 2nd Dose | 12 mg Y14 (B3) | 24 mg Y14 (B3) | 36 mg Y14 (B3) 1st Dose | 36 mg Y14 (B3) 2nd Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng.h/mL | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | 16.4 (83) | NA (NA) — BLQ | 24.4 (21) | 26.3 (105) | 34.0 (50) | 33.4 (51) | NA (NA) — BLQ | NA (NA) — BLQ | 19.7 (89.7) | 53.2 (21) | 76.7 (26) | 89.6 (17) | 81.2 (45) | 10.1 (303) | 38.1 (34) | 82.1 (21) | 63.6 (76) | 9.67 (165) | 40.4 (36) | 86.6 (22) | 87.2 (34)

4. Secondary Outcome: AUC 0-τ
Description: The area under the concentration versus time curve within a (168 h) dosing interval, calculated by the mixed linear/log trapezoidal rule (equivalent to AUC0-168h, which was calculated as the area under the concentration versus time curve from time zero to 168 h post-dose after a single dose, calculated by the mixed linear/log trapezoidal rule).
Time Frame: Up to 168h after dosing
Population: PK Parameters: N/A = For the doses given to cohorts A1, A2, A3 and A4, Y14 was below the LLOQ(<0.2 ng/mL) in most samples (BLQ=below the limit of quantification), so the data for cohort A5 onwards are presented. Only subjects receiving Y14 were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD A2-A9 | Placebo (Part B) | 9 mg Y14 (B1) | 12 mg Y14 (B1) | 16 mg Y14 (B1) | 20 mg Y14 (B1) | 26 mg Y14 (B1) | 9 mg Y14 (B2) | 24 mg Y14 (B2) | 36 mg Y14 (B2) 1st Dose | 36mg Y14 (B2) 2nd Dose | 12 mg Y14 (B3) | 24 mg Y14 (B3) | 36 mg Y14 (B3) 1st Dose | 36 mg Y14 (B3) 2nd Dose
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng.h/mL | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | NA (NA) — BLQ | 64.0 (105) | 164 (199) | 65.2 (126) | 78.2 (47) | 59.2 (84.6) | NA (NA) — BLQ | NA (NA) — BLQ | 24.8 (127) | 108 (18.7) | 139 (17) | 153 (16) | 144 (53) | 15.6 (598) | 107 (31) | 159 (25) | 154 (76) | 17.0 (298) | 106 (28) | 193 (19) | 225 (48)

5. Secondary Outcome: T 1/2
Description: Drug Half-life (t1/2) is defined as the amount of time (hours) required for the drug concentration to be reduced to exactly half its initial concentration or amount in blood.
  The apparent terminal half-life, calculated from Loge 2 / λz:
  For Part A cohorts, it was not possible to estimate an unambiguous Tmax or T1/2 due to the extended PK profile of Y14.
  For Part B cohorts, no individual administered dose half-life data were collected for this outcome, but one half-life value was measured after all doses had been administered and these values were analysed only for the treated-arms that is B1, B2 and B3.
Time Frame: For Part A, Cohorts A3 to A9 - up to 840 hour post dose. For Part B - up to day 70 post 1st dose
Population: PK Parameters:
  NA= Values below the limit of quantification (BLQ) For the doses given to cohorts in Part A, Y14 was below the lower limit of quantification (<0.2 ng/mL) in most samples and it was not possible to estimate an unambiguous Tmax or T1/2 due to the extended PK profile of Y14. Therefore the data for Part B only are presented.
  Participants who received placebo were not assessed for this measure, therefore only subjects receiving Y14 were analysed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Placebo (A1): 0.9 % saline single subcutaneous injection
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | 9.0 mg (A2) | 9 mg (A3) | 9 mg (A4) | 18.0 mg (A5) | 36.0 mg (A6) | 18 mg (A7) | 36 mg (A8) | 36 mg (A9) | Placebo SAD (A2-A9) | Placebo (Part B) | 9-26.0 mg (B1) | 9-36 mg (B2) | 12-36 mg (B3)
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 0 | 0 | 6 | 6 | 6
hours |  | NA (NA) — Not available: Below the limit of quantification (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) | NA (NA) — Not available (BLQ) |  |  | 277 (106) | 294 (46) | 190 (28)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks from participant start date
Description: The safety evaluation will include blood pressure, pulse rate, ECG parameters, clinical laboratory tests (haematology, serum biochemistry, coagulation, urinalysis and urine microscopy).
Arm/Group | Placebo (A1) | 1.0 mg (A1) TP1 | 2.0 mg (A1) TP2 | 6.0 mg (A1) TP3 | Placebo SAD (A2-A9) | 9 mg (A4) | 9 mg (A3) | 9.0 mg (A2) | 18 mg (A7) | 18.0 mg (A5) | 36 mg (A8) | 36.0 mg (A6) | 36 mg (A9) | Placebo (Part B) | 9 mg Y14 (B1) | 9 mg Y14 (B2) | 12 mg Y14 (B1) | 12 mg Y14 (B3) | 16 mg Y14 (B1) | 20 mg Y14 (B1) | 24 mg Y14 (B2) | 24 mg Y14 (B3) | 26 mg Y14 (B1) | 36 mg Y14 (B2) | 36 mg Y14 (B3)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/8 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/8 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 3/3 | 3/8 | 5/5 | 4/5 | 1/5 | 5/5 | 5/5 | 4/5 | 5/5 | 5/5 | 3/6 | 5/6 | 4/6 | 6/6 | 5/6 | 6/6 | 6/6 | 6/6 | 5/6 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (A1) (N=3) | 1.0 mg (A1) TP1 (N=3) | 2.0 mg (A1) TP2 (N=3) | 6.0 mg (A1) TP3 (N=3) | Placebo SAD (A2-A9) (N=8) | 9 mg (A4) (N=5) | 9 mg (A3) (N=5) | 9.0 mg (A2) (N=5) | 18 mg (A7) (N=5) | 18.0 mg (A5) (N=5) | 36 mg (A8) (N=5) | 36.0 mg (A6) (N=5) | 36 mg (A9) (N=5) | Placebo (Part B) (N=6) | 9 mg Y14 (B1) (N=6) | 9 mg Y14 (B2) (N=6) | 12 mg Y14 (B1) (N=6) | 12 mg Y14 (B3) (N=6) | 16 mg Y14 (B1) (N=6) | 20 mg Y14 (B1) (N=6) | 24 mg Y14 (B2) (N=6) | 24 mg Y14 (B3) (N=6) | 26 mg Y14 (B1) (N=6) | 36 mg Y14 (B2) (N=6) | 36 mg Y14 (B3) (N=6)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 4 (5) | 4 (4) | 5 (13) | 3 (3) | 0 (0) | 4 (7) | 1 (2) | 2 (2) | 0 (0) | 4 (5) | 3 (3) | 3 (5) | 1 (1) | 2 (2) | 2 (2) | 3 (4)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early Satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 6 (12)
Injection site injuration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 5 (5) | 5 (5) | 4 (4) | 5 (5) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 4 (4) | 3 (3) | 4 (4) | 5 (5) | 5 (5) | 4 (7) | 6 (11)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 4 (6) | 2 (5)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (5) | 2 (5) | 1 (1) | 2 (2) | 3 (8) | 2 (4) | 3 (4) | 0 (0) | 2 (3) | 2 (4) | 3 (4) | 1 (1) | 3 (4) | 2 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food craving (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03673111/Prot_SAP_000.pdf